In this abbreviated Statistical Analysis Plan (SAP), we present the tables/figures to be produced for TACTILE. We retain the paragraph numbering from the original SAP.

## 8.1 Patient Accountability

The number and percentage of randomized and withdrawn patients will be presented by treatment group (Table 14.1.1). The number and percentage of enrolled patients prematurely discontinuing the study will also be presented by treatment group together with the reason for withdrawal. Patient accountability will also be presented by site stratified by treatment group (Table 14.1.2).

## 8.2 Safety Analyses

Descriptive statistics and appropriate tests will be used to summarize and compare the safety parameters between treatment groups. All safety analyses will be performed on the safety population. Treatment group comparisons will assess the significance of the difference between treatment and control groups.

#### 8.2.1 Adverse Events

Adverse events will be coded according to pre-specified Tactile internal codes. Adverse events will be summarized by severity, outcome, causality and seriousness (i.e., SAE) and stratified by treatment group (Table 14.3.1). For subjects with more than one event, the event with the highest level of severity, outcome or causality, seriousness, respectively, will be reported. The number and percentage of subjects with an event by the internal Tactile AE codes will be compared by treatment group (Tables 14.3.2). Subjects with more than one event by internal Tactile code will be counted only once. All AEs will be listed, sorted by treatment group, subject identification, and date of the AE (Table 16.2.7.1). Data presented will include: causality, severity, seriousness, outcome, verbatim description, internal Tactile codes.

#### 8.2.2 Serious Adverse Events

SAEs will be listed, sorted by treatment group, subject identification, and onset date (Table 16.2.7.2). Data presented will include: causality, severity, seriousness, outcome, verbatim description, internal Tactile codes.

# 8.2.3 Other Safety Analyses

The following analyses will be carried out on the Safety Populations. ACTitouch® treated subjects will be compared with multi-layer bandaging treated subjects in terms of:

the difference in the incidence of ulcer-related adverse events (defined as ulcer infections, maceration, allergic reaction to dressing, or hospitalization for worsening VLU) at 16 weeks using the Cochrane-Mantel-Haenszel (CMH) test (Table 14.3.3).

# 8.3 Efficacy Analyses

All analyses will be carried out on the ITT population.

# 8.3.1 Primary Efficacy Analysis

The percentage of each subject's ulcer area reduction at 16 weeks will be assessed using a specialized ulcer camera and ulcer imaging system. Images will be centrally read by a qualified independent adjudicator. The percentage of ulcer area reduction for the ACTitouch® treated subjects will be compared with multi-layer bandaging treated subjects using a linear mixed model analysis of covariance (ANCOVA) with the following covariates: treatment group; duration of VLU ([1,6]; (6,24] months); baseline size of VLU, [1.5,12cm], (12,50cm]; history of diabetes; age. The analysis will be conducted on the ITT population (Table 14.2.3).

# 8.3.2 Secondary Efficacy Analysis

The following analyses will be carried out on all three analysis populations defined above.:

• ACTitouch® treated subjects will be compared with multi-layer bandaging treated subjects in terms of the difference in changes in HRQOL at 16 weeks assessed by the overall score of the Charing Cross Venous Ulcer Questionnaire using a similar ANCOVA model as used in similar to the Primary Endpoint Analysis. If the primary efficacy analysis was significant, then the difference will be tested at the two-sided α=.05 level – Table 14.2.6.

## 8.3.3 Exploratory Efficacy Analysis

- To compare the difference in ulcer-free days at 16 weeks between ACTitouch® treated subjects with multi-layer bandaging treated subjects based on non-parametric analysis of covariance using the same covariates -Table 14.2.7.
- To compare the difference in changes in HRQOL at 16 weeks compared to baseline between ACTitouch® treated subjects with multi-layer bandaging treated subjects using the overall score of the VCSS and the same method as the Primary Endpoint Analysis -Table 14.2.10
- To compare the difference in the time-to-100% healed VLU between ACTitouch® treated subjects with multi-layer bandages treated subjects using a Cox Proportional Hazard model with the same covariates as above -Table 14.2.12.
- To compare the cumulative incidence graphs of subjects with 100% percent healed VLU between ACTitouch® treated subjects with multi-layer bandaging treated subjects using Kaplan-Meier product-moment estimates and the log rank rest for differences in survival curves - Figure 1.

Accepted: Date: ROCF 2017

Name: Sunday Hoy, Director of Clinical Resources and Research, Tactile Medical

# **APPENDIX: DATA TABLES**

Sponsor: Tactile Medical Systems Protocol: 6010

Table 14.1.1 Patient Disposition ITT sample

page 1 of x

| | | | 1.5cm<=si | ze<=12cm | | | 12cm <size<= 500<="" th=""><th>m</th></size<=> | m |
|---|---|---|---|---|---|---|---|---|
| | 1<=age< | <6 months | 1<=age | <6 months | 6<= | age<=24 months | 6<=a | ge<= 24 months |
| | Treatment<br>(N) | Control<br>(N) | Treatment<br>(N) | Control<br>(N) | Treatment<br>(N) | Control<br>(N) | Treatment (N) | Control<br>(N) |
| Randomized | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) |
| Safety | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) |
| Completed | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) |
| Discontinued | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) |
| Primary Reason for<br>Discontinuation: | | | | | | | | |
| Adverse Event | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) |
| Protocol Violation | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) |
| Lost to Follow-up<br>Other | xx/xx(xxx.x%)<br>xx/xx(xxx.x%) | xx/xx(xxx.x%)<br>xx/xx(xxx.x%) | xx/xx(xxx.x%)<br>xx/xx(xxx.x%) | xx/xx(xxx.x%)<br>xx/xx(xxx.x%) | xx/xx(xxx.x%)<br>xx/xx(xxx.x%) | xx/xx(xxx.x%)<br>xx/xx(xxx.x%) | xx/xx(xxx.x%)<br>xx/xx(xxx.x%) | xx/xx(xxx.x%)<br>xx/xx(xxx.x%) |

Sponsor: Tactile Medical Systems Protocol: 6010

page 1 of x

Table 14.1.2 Patient Disposition By Site ITT sample

| | Treatment N(%) <sup>b</sup> | Control<br>N(%) <sup>b</sup> | Total<br>N(%) <sup>b</sup> |
|---|---|---|---|
| XXXX | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) |
| xxxx | xx/xx(xxx.x%) | xx/xx(xxx.x%) | xx/xx(xxx.x%) |

Note: denominator of all percentages is number randomized by group

Sponsor: Tactile Medical Systems Protocol: 6010


Table 14.3.1 Safety Analysis: Summary Incidence of Adverse Events Safety sample

| Condition | Treatment<br>N(%) | Control<br>N(%) | P-value |
|---|---|---|---|
| Safety Analysis Set | xx | xx | · |
| Patients with Adverse Events | xx(xxx.x%) | xx(xxx.x%) | x.xxx |
| Patients with AEs by Severity <sup>a</sup> | | | |
| No Event | xx(xxx.x%) | xx(xxx.x%) | X.XXX |
| Mild | xx(xxx.x%) | xx(xxx.x%) | |
| Moderate | xx(xxx.x%) | xx(xxx.x%) | |
| Severe | xx(xxx.x%) | xx(xxx.x%) | |
| Patients with AEs by Causality <sup>a</sup> | | | |
| Definitely related | xx(xxx.x%) | xx(xxx.x%) | x.xxx |
| Probably related | xx(xxx.x%) | xx(xxx.x%) | |
| Possibly related | xx(xxx.x%) | xx(xxx.x%) | |
| Not related | xx(xxx.x%) | xx(xxx.x%) | |
| No Event | xx(xxx.x%) | xx(xxx.x%) | |
| Outcome | | | |
| No Event | xx(xxx.x%) | xx(xxx.x%) | x.xxx |
| Resolved | xx(xxx.x%) | xx(xxx.x%) | |
| Resolved w/ sequelae | xx(xxx.x%) | xx(xxx.x%) | |
| Continuing | xx(xxx.x%) | xx(xxx.x%) | |
| Lost to follow-up | xx(xxx.x%) | xx(xxx.x%) | |
| Death | xx(xxx.x%) | xx(xxx.x%) | |

| Condition | Treatment N(%) | Control<br>N(%) | P-value |
|---------------------------------|----------------|-----------------|---------|
| Patients with SAEs | xx(xxx.x%) | xx(xxx.x%) | X.XXX |
| Patients Discontinued due to AE | xx(xxx.x%) | xx(xxx.x%) | x.xxx |

NOTE: P-value based on Kruskal-Wallis test controlling for stratification. Denominator is the number of patients in the Safety Analysis Set. 
<sup>a</sup>Patients experiencing more than one adverse event are counted under the maximum severity experienced across events.

Sponsor: Tactile Medical Systems Protocol: 6010


Table 14.3.2 Safety Analysis: Incidence of Adverse Events by Internal AE Code Safety sample

| Internal AE Code | Treatment N(%) | Control<br>N(%) | p-value <sup>a</sup> |
|---|---|---|---|
| Patients with Adverse Events | xx(xxx.x%) | xx(xxx.x%) | xxxx |
| AE_CODE XX | xx(xxx.x%) | xx(xxx.x%) | x.xxx |

Note: A patient experiencing multiple incidences of an event with the same internal AE code is counted only once.

<sup>a</sup> P-value calculated from CMH Test.

Sponsor: Tactile Medical Systems Protocol: 6010

### Table 16.2.7.1 Listing of Adverse Events Safety sample


| Treatment<br>Group | Patient ID | Onset Date<br>(Study Day) | Stop Date<br>(Study Day) | Internal<br>AE Code | Serious | Duration | Severity | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | xx | ddmmyy (xx) | ddmmyy(xx) | XX | xx | XX | XX | xx | xx |
| xxxx | xx | ddmmyy (xx) | ddmmyy(xx) | xx | xx | xx | xx | xx | xx |
| xxxx | xx | ddmmyy(xx) | ddmmyy(xx) | xx | xx | xx | xx | xx | xx |
| xxx | xx | ddmmyy(xx) | ddmmyy(xx) | xx | xx | xx | xx | xx | xx |
| XXXX | xx | ddmmyy(xx) | ddmmyy(xx) | xx | xx | xx | xx | xx | xx |

Sponsor: Tactile Medical Systems Protocol: 6010


Table 14.3.3 Safety Analysis: Incidence of Ulcer-Related Adverse Events at 16 Weeks
Safety sample

| Ulcer-related AE | Trootmant | Control | n volue |
|---|---|---|---|
| Ulcer-related AE | Treatment | | p-value <sup>a</sup> |
| | N(%) | N(%) | |
| Ulcer infecttions | xx/xx(xxx.x%) | xx/xx(xxx.x%) | x.xxx |
| Ulcer maceration | xx/xx(xxx.x%) | xx/xx(xxx.x%) | x.xxx |
| Allergic reactions | xx/xx(xxx.x%) | xx/xx(xxx.x%) | x.xxx |
| Hospitalization for worsening VLU | xx/xx(xxx.x%) | xx/xx(xxx.x%) | x.xxx |
| All Ulcer-related AEs | xx/xx(xxx.x%) | xx/xx(xxx.x%) | x.xxx |

Note: P-value calculated using the CMH test adjusting for ulcer size and duration (stratification)

Sponsor: Tactile Medical Systems

Protocol: 6010


Table 14.2.3 Primary Efficacy Analysis: Changes in % Wound Area Reduction
Evaluable Available Case Population

| | | % Wound Area Redu | ction at Follow-up | Changes in % Wour<br>from Ba | | | |
|---|---|---|---|---|---|---|---|
| · Label | Statistic | Treatment Group<br>(N=122) | Control Group<br>(N=128) | Treatment Group | Control Group | [Treatment -<br>Control]<br>Difference<br>(95% CI)* | P-Value <sup>£</sup> |
| baseline | N | xx | xx | | | | |
| | Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | | | | |
| | Median(Min,Max) | xx(xx,xx) | xx(xx,xx) | | | | |
| 16 weeks | N | xx | xx | xx | xx | | |
| | Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x( xx.x, xx.x) * | $X.XXX^{\mathfrak{E}}$ |
| | Median(Min,Max) | xx(xx,xx) | xx(xx,xx) | xx(xx,xx) | xx(xx,xx) | | |

NOTES:\* Estimates of mean difference between treatment groups, 95% confidence interval and P-value based on a linear mixed model ANCOVA with the following covariates: treatment group; duration of VLU ([1,6]; (6,24] months); baseline size of VLU, [1.5,12cm], (12,50cm]; history of diabetes; age. \* The covariate adjusted one-sided lower bound 97.5% confidence interval of the treatment difference in mean percent ulcer area reduction (calculated as mean of ACTitouch® group minus mean of multi-layer bandaging treated group) is compared to the non-inferiority margin (-.125) . If the lower bound exceeds the margin, the null hypothesis is rejected, and ACTitouch® system is deemed non-inferior to multi-layer bandaging.

Sponsor: Tactile Medical Systems Protocol: 6010


Table 14.2.6 Secondary Efficacy Analysis: Changes in Charing Cross Scores at 16 Weeks Evaluable Available Case Population

| | | % Wound Area | at Follow-up | Changes in % Wound | Area from Baseline | | |
|---|---|---|---|---|---|---|---|
| Label | Statistic | Treatment Group<br>(N=122) | Control Group<br>(N=128) | Treatment Group | Control Group | [Treatment -<br>Control]<br>Difference<br>(95% Cl)* | P-Value <sup>¥</sup> |
| baseline | N | xx | xx | | | | |
| | Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | | | | |
| | Median(Min,Max) | xx(xx,xx) | XX(XX,XX) | | | | |
| 16 weeks | N | xx | xx | . xx | xx | | |
| | Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x( xx.x, xx.x) | x.xxx |
| | Median(Min,Max) | xx(xx,xx) | xx(xx,xx) | xx(xx,xx) | xx(xx,xx) | | |

Note: \*Estimates of mean difference between treatment groups, 95% confidence interval and P-value based on linear mixed model ANCOVA with the following covariates: treatment group; duration of VLU ([1,6]; (6,24] months); baseline size of VLU, [1.5,12cm], (12,50cm]; history of diabetes; age.

Sponsor: Tactile Medical Systems

Protocol: 6010


Table 14.2.7 Exploratory Efficacy Analysis: Ulcer Free Days at 16 Weeks
Evaluable Available Case Population

| | | % Wound Area | at Follow-up | Changes in % Wound | Area from Baseline | | |
|---|---|---|---|---|---|---|---|
| Label | Statistic | Treatment Group<br>(N=122) | Control Group<br>(N=128) | Treatment Group | Control Group | [Treatment -<br>Control]<br>Difference<br>(95% CI)* | P-Value <sup>¥</sup> |
| baseline | N | XX | xx | | | | |
| | Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | | | | |
| | Median(Min,Max) | xx(xx,xx) | xx(xx,xx) | | | | |
| 16 weeks | N | xx | xx | ×× | xx | | |
| | Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x( xx.x, xx.x) | X.XXX |
| | Median(Min,Max) | xx(xx,xx) | xx(xx,xx) | xx(xx,xx) | xx(xx,xx) | | |

Note: \*Estimates of mean difference between treatment groups, 95% confidence interval and P-value based on non-parametric ANCOVA with the following covariates: treatment group; duration of VLU ([1,6]; (6,24] months); baseline size of VLU, [1.5,12cm], (12,50cm]; history of diabetes; age.

Sponsor: Tactile Medical Systems Protocol: 6010


Table 14.2.10 Exploratory Efficacy Analysis: Changes in VCSS at 16 Weeks Evaluable Available Case Population

| 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | % Wound Area | at Follow-up | Changes in % Wound | Area from Baseline | | |
|---|---|---|---|---|---|---|---|
| Label | Statistic | Treatment Group<br>(N=122) | Control Group<br>(N=128) | Treatment Group | Control Group | [Treatment -<br>Control]<br>Difference<br>(95% CI)¥ | P-Value <sup>¥</sup> |
| baseline | N | xx | xx | | | | |
| | Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | | | | |
| | Median(Min,Max) | xx(xx,xx) | xx(xx,xx) | | | | |
| 16 weeks | N | xx | . <b>xx</b> | xx | xx | | |
| | Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x( xx.x, xx.x) | x.xxx |
| | Median(Min,Max) | xx(xx,xx) | xx(xx,xx) | xx(xx,xx) | xx(xx,xx) | | |

Note: \*Estimates of mean difference between treatment groups, 95% confidence interval and P-value based on ANCOVA with the following covariates: treatment group; duration of VLU ([1,6]; (6,24] months); baseline size of VLU, [1.5,12cm], (12,50cm]; history of diabetes; age.

Sponsor: Tactile Medical Systems Protocol: 6010


Table 14.2.11. Exploratory Analysis: Cox PH Analysis of the Time to 100% Healed VLU

| | | 95% Confidence Interval | |
|-----------------|-------------|-------------------------|---------|
| Variable | Hazard Rate | Hazard Rate | P-value |
| Treatment Group | x.xxx | ( x.xxx, x.xxx) | x.xxx |
| Ulcer Size | x.xxx | ( x.xxx, x.xxx) | x.xxx |
| Jicer Duration | x.xxx | ( x.xxx, x.xxx) | x.xxx |
| Diabetes | x.xxx | ( x.xxx, x.xxx) | x.xxx |
| <b>A</b> ge | X.XXX | ( x.xxx, x.xxx) | x.xxx |